CLINICAL TRIAL: NCT01689298
Title: Carbetocin vs. Oxytocin: In-vitro Myometrial Contractions With and Without Oxytocin Pre-treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-05; 11-0257-E (Other: REB (MSH))
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Dose response; Oxytocin pretreatment; Oxytocin; Carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No drug pre-treatment (Active Comparator): A control sample from each patient (no uterotonic drug will be applied during pre-treatment) will be measured concurrently with samples pre-treated with oxytocin. Controls will undergo the same dose response of oxytocin or carbetocin after pre-treatment period as the groups given oxytocin for pre-treatment.
  Interventions: Drug: Oxytocin; Drug: Carbetocin
- Drug pre-treatment (Active Comparator): A sample from each patient will be pre-treated with oxytocin 10-5mol/L. These samples will undergo the same dose response of oxytocin or carbetocin after pre-treatment period as the groups given no drug for pre-treatment (controls).
  Interventions: Drug: Oxytocin; Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
  Other Names: Pitocin
Drug: Carbetocin — Carbetocin, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
  Other Names: Duratocin

SUMMARY:
The purpose of this study is to compare the ability of an isolated sample of uterine muscle tissue (in a tissue bath) to contract in the presence of various drugs. The drugs studied--uterotonics--are typically used to contract the uterus when a pregnant patient continues to bleed after delivery. Oxytocin is an old standard, but seems to suffer from a desensitization phenomenon. Carbetocin, a similar drug, has recently been suggested to clinicians as a replacement for oxytocin directly after certain types of Cesarean section.

The investigators will be testing isolated uterine muscle samples after pre-treatment with oxytocin OR nothing (control) to increasing concentrations of oxytocin OR carbetocin. Contractile measures will be measured and compared between all groups. The investigators hypothesize that oxytocin pre-treatment will reduce contractions in both oxytocin- and carbetocin-induced contractions, and oxytocin and carbetocin will induce different patterns of contractions.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a major cause of maternal mortality and morbidity. In 80% cases of PPH, the primary cause is failure of the uterus to contract after delivery of the baby, which then requires further treatment of the mother with uterotonic drugs (drugs used to contract uterus and thus prevent bleeding).

Patients participating in this study will be asked to donate a very small sample of uterine tissue during Cesarean section, which will be tested in the laboratory for the ability to contract in response to the uterotonics oxytocin and carbetocin. We will seek to better understand the effects of these drugs by comparing their contractile capability in isolated uterine tissue.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary or first repeat Cesarean section
* Cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who require general anesthesia
* Patient who had previous myometrial surgery or more than one previous Cesarean section
* Patients with placental anomalies
* Emergency Cesarean section in labor
* Patients with multiple pregnancy (twins, etc.)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Amplitude of contraction | 6-8 hours

SECONDARY OUTCOMES:
Integrated area under response curve (AUC) | 6-8 hours
Basal tone | 6-8 hours
Frequency of contraction | 6-8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada